CLINICAL TRIAL: NCT01047592
Title: N-methyl-D-aspartate (NMDA) Enhancers' Benefit to Schizophrenia Treatment
Brief Title: Treatment of N-methyl-D-aspartate (NMDA) Enhancers for Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang-Hua Hospital (Other Government)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chun Yuan Lin , MD, Attending, Chang-Hua Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR98-IR-014; HAC9814 (Other: Hospital Adminstration Comission, DOH, Taiwan)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; cognitive function; N-methyl-D-aspartate receptor
MeSH Terms: conditions — Schizophrenia | interventions — Sarcosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sarcosine (Active Comparator)
  Interventions: Drug: sarcosine
- sarcosine+ BE (Active Comparator)
  Interventions: Drug: sarcosine+ BE
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sarcosine — sarcosine, 2 g/d , oral, for 12 weeks
  Arms: sarcosine
Drug: sarcosine+ BE — sarcosine(2 g/d) + BE (1 g/d ), oral, for 12 weeks
  Arms: sarcosine+ BE
Drug: placebo — placebo,oral, for 12 weeks
  Arms: Placebo

SUMMARY:
Hypofunction of N-methyl-D-aspartate (NMDA) receptor has been implicated in the pathophysiology of schizophrenia. To date, several reported trials on adjuvant NMDA-enhancing agents, including glycine and sarcosine (a glycine transporter I inhibitor), demonstrated clinical benefits for schizophrenia patients. This project aims to compare the efficacy and safety of sarcosine and combination of sarcosine and BE, as adjunctive therapy for schizophrenia, and to explore the possible synergistic effects of them. Sixty chronic schizophrenic inpatients will be enrolled in the 12-week double-blind, placebo-controlled trial. The participants receive stable antipsychotic regimens concomitant with sarcosine (2 g/d) (N=21), sarcosine(2 g/d) + BE(1 g/d ) (N=21), and placebo(N=21). Measures of clinical efficacy and side-effects were determined every 3 weeks. Measures of cognitive function were determined at the beginning and the end of the study. The efficacies of three groups are compared, and the characteristics of better responders are analyzed.

DETAILED DESCRIPTION:
We will measure clinical efficacy every 3 weeks during the treatment. At the beginning and the end of the trial,We will utilize a battery of tests to assess the effect of the treatment on cognitive functions.The side effect assessments are also performed every 3 weeks. Side effect assessments include Simpson-Angus Rating Scale for extrapyramidal side-effects, Abnormal Involuntary Movement Scale (AIMS) for dyskinesia, and Barnes Akathisia Scale. Systemic side effects are reviewed by applying the Udvalg for Kliniske Undersogelser (UKU) Side-effects Rating Scale. DAAO level, routine laboratory tests, including CBC, biochemistry , urine analysis, and EKG, will be checked at baseline and the end of week 12.

To compare the metabolic syndrome parameters among groups, body mass index, hip size, waist size, blood pressure, fasting blood sugar, triglyceride, and total-cholesterol will be checked at baseline and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The participants fulfill the criteria of schizophrenia according to the
* Diagnostic and Statistic Manual, fourth edition (DSM-IV).
* The participants remain stable schizophrenic symptoms and receive stable antipsychotic regimens at last 8 weeks before enrollment.
* The participants agree to participate in the study and provide informed consent.

Exclusion Criteria:

* History of alcohol or substance dependence, history of epilepsy, head trauma or CNS diseases, history of major, untreated medical diseases, mental retardation, pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Positive, negative, cognitive symptoms of schizophrenia, laboratory tests. | 12 weeks

SECONDARY OUTCOMES:
The subscales of PANSS,MATRICS, and serum DAAO levels. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chun-yuan Lin, MD, Principal Investigator — Changhua Hospital; Hsien-yuan Lane, MD,PHD, Study Director — China Medical University Hospital
Locations (1):
- Changhua Hospital, Changhua, Taiwan, Taiwan